CLINICAL TRIAL: NCT05477836
Title: Feasibility and Safety of MiWEndo-assisted Colonoscopy:Pilot Study
Brief Title: Feasibility and Safety of MiWEndo-assisted Colonoscopy
Acronym: MiWEndo1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiWEndo Solutions S.L. (Industry)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DO-021_CIP1
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Colorectal Neoplasms; Colorectal Adenomatous Polyp; Colorectal Adenocarcinoma
Keywords: microwave imaging; colonoscopy; early diagnosis; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Traditional feasibility study, following a single-center prospective, non-comparative, with few patients design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Microwave-based colonoscopy
  Interventions: Device: MiWEndo-assisted colonoscopy

INTERVENTIONS:
Device: MiWEndo-assisted colonoscopy — All colonoscopies will be performed with high-definition technology. The MiWEndo System (MiWEndo Solutions, Barcelona) will be fitted to the tip of the endoscope before colonoscopy is started and connected to the microwave processor unit. Endoscopies will be performed by experienced endoscopists who will be previously trained on the use of the MiWEndo System.
  At the beginning of the extubation, the MiWEndo System will be turned on. During extubation, each segment will be carefully examined with both white light and MiWEndo. In case one of them identifies a polyp, the exploration will be stopped and check if it has been detected by the alternative method as well. All the polyps will be resected and sent to the Pathological Department for histological analysis following the usual clinical practice. A stopwatch will be used to measure both total procedure time and withdrawal time.

SUMMARY:
The study involves the planned use of a new microwave-based device during colonoscopy procedures in a small group of patients to assess the preliminary safety of its use and lack of normal clinical practice modification. The device is a final design version, which has been previously tested in several preclinical studies, including: phantom studies, an ex vivo study with human tissues, and an in vivo study with animal model (pig).

DETAILED DESCRIPTION:
This study is designed as a single-center prospective, non-comparative, first in human pilot safety and feasibility study with few patients, whereby data will be subject to an analytical description, rather than to a statistical treatment (refer to Statistical design and analysis).

In this study the principal aim is to assess the clinical safety of the device and the feasibility of its use in assisted colonoscopy. Relevant claims to verify in this study are that the device can be used without ADEs, without any change in the current clinical practice, as well as without any major difficulty by the endoscopist, neither in the preparation nor in the use of the device during exploration.

In addition, the study aims to gather real clinical data with the use of the device to optimise the processing software that will be key to demonstrate MiWEndo's performance on a subsequent clinical investigation (pivotal study).

Consequently, principal and secondary objectives of this investigation, are:

* Principal objectives:

  * To assess the feasibility of performing a complete colonoscopy using the MiWEndo System.
  * To assess the safety of MiWEndo colonoscopy.
* Secondary objectives:

  * To assess the perception of difficulty by the endoscopist when the device is used.
  * To assess the patient's comfort.
  * To collect data on polyp detection performance to guide possible further improvements of the software before starting the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 50 years referred for a diagnostic or surveillance colonoscopy and having signed the Informed Consent Form.

Exclusion Criteria:

* Patients at a high risk of having major complications as perforation or hemorrhage or in whom the possibility of performing a complete colonoscopy is reduced, including: patients with known colonic strictures, total colectomy, acute diverticulitis, inflammatory bowel disease, suspected or proven lower gastrointestinal bleeding, non-correctable coagulopathy or anticoagulant/clopidogrel therapy during procedure, inadequate bowel cleansing or previous incomplete colonoscopy.
* ASA-IV patients
* Urgent colonoscopy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Number of incidents and adverse events | During the procedure and up to 2 weeks after
  To assess the safety of MiWEndo colonoscopy using the lexicon proposed by the American Society of Gastrointestinal Endoscopy (ASGE).
Number of mural injuries | During the procedure
  To assess the safety of MiWEndo colonoscopy according to the Sydney classification for deep mural injuries (DMI)
Rate of cecal intubation | During the procedure
  To assess the feasibility of performing a complete colonoscopy using the MiWEndo System. This parameter will be measured as complete colonoscopy (yes/no).
Length of colon explored | During the procedure
  In case cecum could not be reached, the distance will be measured (in cm).

SECONDARY OUTCOMES:
Patients' comfort | Immediately after the procedure and 2 weeks after
  Subjective assessment from patient following the Gloucester 5-Likert scale, where 1 is no discomfort and 5 is extreme discomfort.
Time for reaching the cecum (or maximum explored colon length) | During the procedure
  Measured in minutes
Total time for completing the procedure | Immediately after the procedure
  Measured in minutes
Perception of difficulty | Immediately after the procedure
  Difficulty by the endoscopist subjectively assessed based on a 5-points Likert scale, where 0 is not difficult and 4 is very difficult.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No